CLINICAL TRIAL: NCT03787602
Title: A Phase 1b/2, Open-Label Study Evaluating the Safety and Efficacy of KRT-232 in Patients With p53 Wild-Type (p53WT) Merkel Cell Carcinoma (MCC) Who Have Failed Anti-PD-1 or Anti-PD-L1 Immunotherapy, or in Combination With Avelumab in MCC Patients Who Are Anti-PD-1 or Anti-PD-L1 Treatment Naïve
Brief Title: Navtemadlin (KRT-232) With or Without Anti-PD-1/Anti-PD-L1 for the Treatment of Patients With Merkel Cell Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kartos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRT-232-103
Record Dates: First submitted 2018-12-06; First posted 2018-12-26 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Merkel Cell Carcinoma
Keywords: navtemadlin (KRT-232)
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Cohort 1, Arm 1 (Experimental): KRT-232 will be administered orally, once daily (QD) on Days 1-7 in a 21-day cycle.
  Interventions: Drug: KRT-232
- Cohort 1, Arm 1b (Experimental): KRT-232 will be administered orally, once daily (QD) on Days 1-5 in a 23-day cycle.
  Interventions: Drug: KRT-232
- Cohort 1, Arm 2b (Experimental): KRT-232 will be administered orally, once daily (QD) on Days 1-5 in a 28-day cycle.
  Interventions: Drug: KRT-232
- Cohort 1, Arm 3 (Experimental): KRT-232 will be administered orally, once daily (QD) on Days 1-7 in a 21-day cycle.
  Interventions: Drug: KRT-232
- Cohort 1, Arm 5 (Experimental): KRT-232 will be administered orally, once daily (QD) on Days 1-7 in a 28-day cycle.
  Interventions: Drug: KRT-232
- Cohort 1 Expansion (Experimental): KRT-232 will be administered orally, once daily (QD) per Cohort 1 RP2D dose and schedule.
  Interventions: Drug: KRT-232
- Cohort 2, Arm 1 KRT-232 in combination with avelumab (Experimental): KRT-232 will be administered orally, once daily (QD) on Days 1-5, in combination with avelumab 800 mg IV on Day 1 and 15 in a 28-day cycle.
  Interventions: Drug: KRT-232; Drug: Avelumab
- Cohort 2, Arm 2 KRT-232 in combination with avelumab (Experimental): KRT-232 will be administered orally, once daily (QD) on Days 1-7, in combination with avelumab 800 mg IV on Day 1 and 15 in a 28-day cycle.
  Interventions: Drug: KRT-232; Drug: Avelumab
- Cohort 2 Expansion (Experimental): KRT-232 will be administered orally, once daily (QD) per RP2D dose and schedule, in combination with avelumab 800 mg IV on Day 1 and 15 in a 28-day cycle.
  Interventions: Drug: KRT-232; Drug: Avelumab
- Cohort 3 (Experimental): KRT-232 will be administered orally, once daily (QD) per Cohort 1 RP2D dose and schedule.
  Interventions: Drug: KRT-232
- Cohort 4 (Experimental): KRT-232 will be administered orally, once daily (QD) per Cohort 1 RP2D dose and schedule.
  Interventions: Drug: KRT-232

INTERVENTIONS:
Drug: KRT-232 — KRT-232 is an experimental MDM2 anticancer drug taken by mouth.
  Other Names: navtemadlin
Drug: Avelumab — Avelumab is a PD-L1 blocking antibody anticancer drug administered by intravenous infusion.
  Other Names: Bavencio
  Arms: Cohort 2 Expansion; Cohort 2, Arm 1 KRT-232 in combination with avelumab; Cohort 2, Arm 2 KRT-232 in combination with avelumab

SUMMARY:
This study evaluates KRT-232, a novel oral small molecule inhibitor of MDM2, for the treatment of patients with Merkel Cell Carcinoma (MCC) who have failed treatment with at least one anti-PD-1 or anti-PD-L1 immunotherapy or in combination with avelumab in MCC patients who are anti-PD-1 or anti-PD-L1 treatment naïve. Inhibition of MDM2 is a novel mechanism of action in MCC.

ELIGIBILITY:
Inclusion Criteria:

* For Cohort 1, 3 and 4 patients must have failed treatment with at least one PD-1 inhibitor or PD-L1 inhibitor for metastatic MCC
* For Cohort 2, patients must not have received any anti-PD-1 or anti-PD-L1 therapy
* For Cohort 3, patients must not have received any prior chemotherapy
* For Cohort 4, patients must have received at least one prior line of chemotherapy
* ECOG performance status of 0 to 1
* Histologically confirmed MCC. Disease must be measurable, with at least 1 measurable lesion by RECIST 1.1
* MCC expressing p53WT based on any CLIA or test approved by local health authority or a validated test (Cohort 1 and 2)
* MCC expressing p53WT based Central Lab test (Cohort 3 and 4)
* Adequate hematological, hepatic, and renal functions

Exclusion Criteria:

* For Cohort 2, subjects must not have autoimmune disease, medical conditions requiring systemic immunosuppression, prior stem cell transplant, or active infection with HBV or HCV.
* Patients previously treated with MDM2 antagonist therapies or p53-directed therapies
* History of major organ transplant
* Patients with known central nervous system (CNS) metastases that are previously untreated
* Grade 2 or higher QTc prolongation (>480 milli-seconds per NCI-CTCAE criteria, version 5.0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Cohort 1 Part 1: To determine the KRT-232 RP2D. | 10 Weeks
  The Safety Review Committee (SRC) will determine RP2D for expansion based on safety and tolerability of each arm.
Cohort 1 Part 2: To determine the objective response rate (ORR) in subjects with p53WT MCC who have failed anti-PD-1 or anti-PDL-1 immunotherapy | 10 Weeks
  ORR will be assessed per RECIST criteria version 1.1 after all subjects have been treated at the RP2D of KRT 232 and completed the second response assessment.
Cohort 2 Part 1: To determine the KRT-232 RP2D in combination with avelumab | 28 Days
  DLTs will be used to establish the MTD of KRT-232 in combination with avelumab. SRC will determine the RP2D based on the safety of combination of KRT-232 with avelumab.
Cohort 2 Part 2: To determine the objective response rate (ORR) in treatment-naïve subjects with p53WT MCC | 10 Weeks
  ORR will be assessed per RECIST criteria version 1.1 after all 30 subjects have been treated at the RP2D of in combination with avelumab and have completed the second response assessment.
Cohort 3: To determine the confirmed overall response rate (ORR) based on IRC assessments in subjects with p53WT MCC are chemotherapy naive and have failed anti-PD-1/PD-L. | 10 Weeks
  ORR will be assessed per RECIST criteria 1.1 by IRC.
Cohort 4: To determine the confirmed overall response rate (ORR) based on IRC assessments in subjects with p53WT MCC who have failed anti-PD-1 or anti-PDL-1 immunotherapy and have had least 1 line of prior chemotherapy. | 10 Weeks
  ORR will be assessed per RECIST criteria 1.1 by IRC.

SECONDARY OUTCOMES:
To determine the confirmed ORR based on investigator assessment. | 1 year after last subject enrolled.
  ORR will be assessed per RECIST criteria 1.1 by investigators.
To determine the duration of response (DoR) | 1 year after last subject enrolled
  Time from documentation of response (CR or PR as determined by RECIST 1.1) until disease progression.
To determine Progression-free survival (PFS) | 1 year after last subject enrolled
  Time from initial treatment until disease progression.
To determine overall survival (OS) | 1 year after last subject enrolled
  Time from initial treatment until death from any cause.
To determine clinical benefit rate (CBR) | 1 year after last subject enrolled.
  PR, CR or stable disease that last at least 10 weeks, per IRC or investigator assessment.

CONTACTS AND LOCATIONS:
Locations (51):
- United States (14):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Miami Cancer Institute, Miami, Florida
  - Moffitt, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Norton Healthcare, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson, Houston, Texas
  - Inova Health Care Services, Fairfax, Virginia
- Princess Alexandra Hospital Oncology, Woolloongabba, Australia
- Brazil (6):
  - Centro Catarinense de Pesquisa (CECAP) - Hospital Santa Catarina de Blumenau, Blumenau
  - Instituto Nacional do Cancer, Brasília
  - Centro Intergado de Oncologia, Curitiba
  - Centro de Pesquisa Clinica em Oncologia, Ijuí
  - Clinica De Neoplasias Litoral, Itajaí
  - Hospital Paulistano, São Paulo
- Princess Margaret Cancer Centre, Toronto, Canada
- France (9):
  - CHU de Bordeaux- Hopital Saint-Andre, Bordeaux
  - AP-HP Universite Paris Saclay, Gif-sur-Yvette
  - CHU de Lille, Lille
  - CHU Lyon-Sud, Lyon
  - Hôpital de la Timone. Aix-Marseille Université, Marseille
  - CHU Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - Hôpital Saint Louis - APHP, Paris
  - CHU de Tours, Tours
- Germany (7):
  - Vivantes Network for Health Gmb, Neukölln Clinic, Berlin
  - Uniklinik Koln, Cologne
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen (AöR), Essen
  - Nationales Centrum für Tumorerkrankungen NCT, Heidelberg
  - Universitätsklinik Rostock, Rostock
  - Universitats-Hautklinik Tubingen, Tübingen
- Italy (5):
  - Institute for Cancer Research and Treatment, Candiolo
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - AUSL della Romagna, Ravenna
  - AOUS Le Scotte, Siena
  - OSP Civile Maggiore Borgo Trento, Verona
- University Medical Center Groningen, Groningen, Netherlands
- South Korea (3):
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (4):
  - Hospital Duran i Reynals, Barcelona
  - Hospital General Universitario Gregorio Marañn (Madrid), Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - Fundacio Investigao Hospital General Universitario de Valencia, Valencia